CLINICAL TRIAL: NCT01189123
Title: Evaluation of Cell-mediated Immunity and Antibody Response to Influenza Vaccination and Correlates of Protection in Seniors
Brief Title: Cell Mediated Immunity in Older Adults
Acronym: CMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Keipp Talbot, Assistant Professor, Infectious Diseases, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 080925; 5U18IP000184-03 (NIH)
Record Dates: First submitted 2010-08-23; First posted 2010-08-26 (Estimated); Results first posted 2014-03-03 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-03

CONDITIONS: Immunity to Influenza Vaccine
Keywords: influenza; vaccine; cell mediated immunity; elderly; high dose influenza vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard dose influenza vaccine (Active Comparator): Fluzone (Sanofi Pasteur)
  Interventions: Biological: fluzone by sanofi pasteur
- High Dose Vaccine (Active Comparator): High Dose Fluzone by sanofi pasteur
  Interventions: Biological: High dose influenza vaccine Sanofi-Pasteur

INTERVENTIONS:
Biological: High dose influenza vaccine Sanofi-Pasteur — High dose influenza vaccine Sanofi-Pasteur at standard dosing intramuscular injection
  Other Names: High dose fluzone (Sanofi-Pasteur)
  Arms: High Dose Vaccine
Biological: fluzone by sanofi pasteur — standard dose fluzone
  Arms: Standard dose influenza vaccine

SUMMARY:
This study is to study the immune response to the flu vaccine in people 65 years old and older. Only adults 65 years old and older and who are getting their flu vaccine are being asked to join in this study. The investigators plan to enroll approximately 100 people in this study in the 2010-2011 flu season. Vanderbilt is working with the Centers for Disease Control and Prevention on this study.

There will be 5 study visits. Up to 4 tablespoons of blood from a vein will be obtained prior to the flu shot. Return visits will be 1, 2, and 4 weeks later,with up to 4 tablespoons of blood drawn again. Patients will be randomized to receive either the standard dose or the high dose flu vaccine. Both flu vaccines are FDA-approved.

DETAILED DESCRIPTION:
During the 2010-2011 influenza season, approximately 100 adults ≥65 years of age will be enrolled. After consent, blood and serum will be collected and then subjects will be randomized to either standard or high dose influenza vaccine (both FDA approved vaccines). Vaccination will be done by an unblinded nurse. All further evaluations and analysis will be done by a blinded staff member. Medical history, relevant medications, and functional/nutritional status will be assessed at the first visit. Subjects will return (Table 3) for blood and serum draws on days 7, 14, 28 and for a serum blood draw after influenza season. No micronutrient samples will be drawn, but serum will be kept for possible vitamin D testing. During influenza season, subjects will answer a questionnaire about influenza-like illness (ILI) every two weeks (either by email or telephone) and will be asked to return for a nasal swab if an ILI is present. Comparisons will be made of the cell-mediated response of those vaccinated with standard versus high dose vaccines. Analyses will be done accounting for age, use of immunomodulating agents, and underlying medical conditions.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* aged 65+ years

Exclusion Criteria:

* <65 years
* influenza vaccine allergy
* Guillain-Barre
* weight <110 pounds

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 105 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. Keipp Talbot, MD MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Kim JH, Talbot HK, Mishina M, Zhu Y, Chen J, Cao W, Reber AJ, Griffin MR, Shay DK, Spencer SM, Sambhara S. High-dose influenza vaccine favors acute plasmablast responses rather than long-term cellular responses. Vaccine. 2016 Aug 31;34(38):4594-4601. doi: 10.1016/j.vaccine.2016.07.018. Epub 2016 Jul 26. PMID 27473306

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Dose Influenza Vaccine: Fluzone (Sanofi Pasteur)
  fluzone by sanofi pasteur: standard dose fluzone
  1 dose of vaccine was given IM
- High Dose Vaccine: High Dose Fluzone by sanofi pasteur
  High dose influenza vaccine Sanofi-Pasteur: High dose influenza vaccine Sanofi-Pasteur at standard dosing (1 IM injection)
Period: Overall Study
Arm/Group | Standard Dose Influenza Vaccine | High Dose Vaccine
Started | 52 | 53
Completed | 50 | 47
Not Completed | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Dose Influenza Vaccine | High Dose Vaccine | Total
Number analyzed (Participants) | 52 | 53 | 105
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 74 [68 to 77] | 72 [67 to 79] | 73 [67 to 77]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 52 | 53 | 105
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 51
  Male | 27 | 27 | 54
Region of Enrollment [Number; unit: participants]
  United States | 52 | 53 | 105

OUTCOME MEASURES:

1. Primary Outcome: Cellular Immune Response
Description: comparison of CMI in high vs standard dose
Time Frame: 3 years
Population: A subset of samples were chosen for testing since not enough money was available to test samples from all subjects. The samples were divided by randomization group (blinded to study staff -- they were called group A or group B). From each group, samples were randomly pulled.
Measure: Median (Inter-Quartile Range); unit: percentage of Stimulated cells
Arm/Group | Standard Dose Influenza Vaccine | High Dose Vaccine
Number analyzed (Participants) | 22 | 26
percentage of Stimulated cells
  CD4+ IFNgamma at Visit 4 | 0.239 [0.124 to 0.396] | 0.137 [0.098 to 0.200]
  CD4+ TNF alpha Visit 4 | 0.243 [0.138 to 0.413] | 0.160 [0.107 to 0.221]
  CD4+ IL2 Visit 4 | 0.174 [0.107 to 0.260] | 0.147 [0.124 to 0.192]
  CD8+ IFNgamma at Visit 4 | 0.162 [0.101 to 0.311] | 0.191 [0.130 to 0.324]
  CD8+ TNF alpha Visit 4 | 0.344 [0.163 to 0.472] | 0.277 [0.126 to 0.485]
  CD8+ IL2 Visit 4 | 0.200 [0.107 to 0.276] | 0.167 [0.108 to 0.289]

2. Secondary Outcome: Antibody Responses
Description: Hemagglutination inhibition antibody titers measured for standard vs high dose
Time Frame: 2 years
Measure: Geometric Mean (95% Confidence Interval); unit: GMT
Arm/Group | Standard Dose Influenza Vaccine | High Dose Vaccine
Number analyzed (Participants) | 50 | 47
GMT
  H1N1 | 40 [10 to 80] | 80 [40 to 160]
  H3N2 | 20 [20 to 40] | 80 [40 to 160]
  B | 40 [20 to 80] | 40 [40 to 80]

ADVERSE EVENTS:
Arm/Group | Standard Dose Influenza Vaccine | High Dose Vaccine
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/53
Other Adverse Events (participants affected / at risk) | 0/52 | 0/53

LIMITATIONS AND CAVEATS:
Due to cost and time limitations, a random sample from each treatment group were pulled for CMI testing. Hence not all samples were tested.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No